CLINICAL TRIAL: NCT01627145
Title: Post-treatment Normallized Urodynamic Findings as the Golden Standard of Objective Cure for Female Overactive Bladder Patients Receiving Antimuscarinic Drug and Its Correlations With Voiding Diary, King's Health Questionnaire, and Overactive Bladder Sympto
Brief Title: Post-treatment Novmalized Urodynamiz Findings as the Golden Standard of Objective Cure for Female Overactive Bladder Patients Receiving Antimuscarinic Drug
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Professor, Department of Obstetrics & Gynecology, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201012024RC
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Overactive Bladder Syndrome
Keywords: overactive bladder syndrome; derusor overactivity; urodynamic studies; bladder oversensitivity
MeSH Terms: interventions — Solifenacin Succinate

ARMS (1):
- antimuscariniz drug (Experimental)
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Solifenacin 5 mg qd,

SUMMARY:
Post-treatment Novmalized Urodynamiz Findings as the Golden Standard of Objective Cure for Female Overactive Bladder Patients Receiving Antimuscarinic Drug and Its Conelations With Voiding Diary, King's Health Quentionaire, Overactive Bladder Sympton Scores and Patient Perception of Bladder Condition.

ELIGIBILITY:
Inclusion Criteria:

* female patients within 18 years old to 99 years old with overactive bladder syndrome

Exclusion Criteria:

* unwilling or unable to perform testing procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of normalized urodynamic pattern after treatment | 12 weeks

SECONDARY OUTCOMES:
The percentage of recurrence rates after treatment during follow-up and further to analyze the risk factors of recurrence | 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- No 8, Chung-Shan South Road,, Taipei, Taiwan, Taiwan